CLINICAL TRIAL: NCT01787643
Title: Adoption of Standing Behavior After Installation of Height-Adjustable Desks
Brief Title: Standing Behavior After Installation of Height-Adjustable Desks
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: USDA Grand Forks Human Nutrition Research Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: GFHNRC702
Record Dates: First submitted 2013-02-06; First posted 2013-02-08 (Estimated); Last update posted 2022-02-02 (Actual); Status verified 2022-01

CONDITIONS: Office Workers; Sitting Occupations
Keywords: height-adjustable desk; office workers; sitting occupations; energy expenditure; BMI; Weight; Lower fat diet
MeSH Terms: conditions — Body Weight | interventions — Working Conditions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Standing desk (Experimental): Installation of standing desk
  Interventions: Other: Height-Adjustable Desk Intallation in Office

INTERVENTIONS:
Other: Height-Adjustable Desk Intallation in Office

SUMMARY:
The purpose of this research study is to determine whether height-adjustable desks change sitting and standing time at work and away from work, engery expenditure, dietary intake, and body composition. Intermittent peroids of standing made possible by height-adjustable desks may help to impart long-term health benefits.

ELIGIBILITY:
Inclusion Criteria:

* Being one of the 18 scientists and support staff who have sedentary jobs
* Voluntarily make the choice to replace their current fixed-height sitting desk for a sit-to-stand height-adjustable desk
* Consents to study conditions

Exclusion Criteria:

* Cannot stand for any type of health of orthopedic reasons
* Do not work fulltime
* Pregnant at baseline or become pregnant during the study

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2013-01; Primary Completion 2014-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Workplace sitting time to be reduced | 12 months
  Workplace sitting time will be reduced by 60 minutes across an 8 hour work day and this time will be replaced by standing.

SECONDARY OUTCOMES:
Total sitting time will be reduced | 12 months
  Total sitting time will be reduced by 30 minutes across a 16 hour day. Decreased sitting during the weekday will not be fully compensated for by increased sitting during nonwork hours.
Energy expenditure will increase | 12 months
  Energy expenditure will increase across an 8 hour workday and a 16 hour day.
Health behavior change of consuming a lower fat diet | 12 months
  The non-targeted health behavior of consuming a lower fat diet will co-occur with standing behavior. Increases in standing behavior will be inversely correlated with changes in total dietary fat intake.
Body weight, BMI, and fat mass reduction | 6 months
  Body weight, BMI, and fast mass will be reduced by 6 months.
Changes in musculoskeletal symptoms | 12 months
  Increases in standing behavior will be correlated with changes in musculoskeletal symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: James Roemmich, PhD, Principal Investigator — USDA Grand Forks Human Nutrition Research Center
Locations (1):
- USDA Grand Forks Human Nutrition Research Center, Grand Forks, North Dakota, United States

REFERENCES:
- [Derived] Roemmich JN. Height-Adjustable Desks: Energy Expenditure, Liking, and Preference of Sitting and Standing. J Phys Act Health. 2016 Oct;13(10):1094-1099. doi: 10.1123/jpah.2015-0397. Epub 2016 Aug 16. PMID 27256708